CLINICAL TRIAL: NCT02704845
Title: Biopsychosocial Exploration of Pain Profiles in Inflammatory and Chronic Non-specific Axial Low Back Pain: An Exploration of Similarities and Differences
Brief Title: Biopsychosocial Exploration of Pain Profiles in Inflammatory and Chronic Non-specific Axial Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Lolwah Al-Rashed, Lead Investigator, University of Dublin, Trinity College
Other Study IDs: UDublinTC 12
Record Dates: First submitted 2016-02-27; First posted 2016-03-10 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Back Pain; Spondylitis, Ankylosing; Low Back Pain
Keywords: Inflammatory back pain; Ankylosing spondylitis; Non-specific low back pain; Pain experience; Disability; Behavioural; Psychological; Biopsychosocial; Pain profiles
MeSH Terms: conditions — Back Pain; Spondylitis, Ankylosing; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Ankylosing Spondylitis
- Chronic non-specific low back pain

SUMMARY:
The biopsychosocial model is well established in chronic low back pain (CLBP) research. Nevertheless, researchers to date have overlooked the biopsychosocial aspects of Inflammatory Low Back pain (ILBP). Most health care providers are biologically oriented in their treatment of ILBP, neglecting its possible multidimensional nature. It is true that people with ILBP may present with more complex pain and physical limitations than those with chronic non-specific low back pain (CNSLBP), but it remains unexplored whether or not these limitations are affected by the same pain factors that affect CNSLBP patients. This study aims to explore and compare the biopsychosocial back pain profiles of adults with ILBP and CNSLBP.

DETAILED DESCRIPTION:
This is a multicentre case-control study that will compare back pain in patients with ankylosing spondylitis and CNSLBP. A multidimensional pain assessment will be conducted for patients in both groups. Each patient will be assessed on one occasion by the same experienced physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 65 years of age
* Low back pain >3 months
* On stable medication
* Ability to walk independently without an assistive device
* Specific inclusion criteria for AS group: clinical diagnosis of ankylosing spondylitis by a rheumatologist
* Specific inclusion for CNSLBP group: clinical diagnosis by a physician for CLBP

Exclusion Criteria:

* Spinal surgery or compression fracture within the last 6 months
* Cauda equine and conus medullaris syndromes
* Severe musculoskeletal conditions affecting the upper and/or the lower limbs, such as severe inflammatory arthritis of the peripheral joints
* Severe osteoporosis
* Leg-length discrepancy
* Cancer
* Morbid obesity, or pregnancy
* Progressive neurological disease
* Psychiatric disease and/or cognitive limitations that could affect the ability to complete the study questionnaires
* Inability to read and/or understand the English language
* Severe cardiac, respiratory or neurological diseases
* Uncontrolled epilepsy
* Specific exclusion criteria for CNSLBP group: Spondyloarthropathy, or any structural abnormalities in the lumbar spine that result in serious neurological dysfunction, such as stage III-IV lumbar disc herniation, and grade III-IV spondylolisthesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of adults with Ankylosing Spondylitis (AS) will be consecutively recruited from a pool of patients referred to AS clinic in the Rheumatology and Physiotherapy Departments of St. James's and Tallaght Hospitals in Dublin.
  Adults with chronic non-specifi low back pain (CNSLBP) (control group) will be consecutively recruited from a pool of patients referred to the Physiotherapy Department of St. James's and Tallaght Hospitals in Dublin. An invitation to participate in the study and an information leaflet will be extended to the patients who potentially meet the recruitment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Back pain intensity - total | Day 1, no follow-up will be required.
  The average total back pain intensity in the last week will be measured by the Numeric Rating Scale (NRS)
Back pain-related functional disability | Day 1, no follow-up will be required.
  Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Back pain beliefs | Day 1, no follow-up will be required.
  Back Beliefs Questionnaire (BBQ)
Pain-related fear, fear of movement/(re)injury | Day 1, no follow-up will be required.
  Tampa Scale for Kinesiophobia (TSK)
The fear-avoidance behaviours of physical activity | Day 1, no follow-up will be required.
  modified Fear Avoidance Behaviour Questionnaire (mFABQ)
Pain catastrophizing behavior | Day 1, no follow-up will be required.
  Pain catastrophizing scale (PCS)
Self-efficacy for AS patients | Day 1, no follow-up will be required.
  Ankylosing Spondylitis-specific Arthritis Self-Efficacy Scale (ASES-AS)
Pain cognition and coping | Day 1, no follow-up will be required.
  Pain Coping Inventory (PCI)
Psychological distress (depression & anxiety) | Day 1, no follow-up will be required.
  Hospital Anxiety and Depression Scale (HADS)
The extent and location of pain | Day 1, no follow-up will be required.
  Pain drawings will be completed for NSCLBP patients on a digital tablet (iPad 2, Apple Computer, Cupertino, CA, USA) using a commercially available sketching software (SketchBook)
Back pain intensity - nocturnal | Day 1, no follow-up will be required.
  The average nocturnal back pain intensity in the last week will be measured by the Numeric Rating Scale (NRS)
Physical function for AS patients | Day 1, no follow-up will be required.
  Bath Ankylosing Spondylitis Functional Index (BASFI)
Disease activity for AS patients | Day 1, no follow-up will be required.
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Disease activity for AS patients | Day 1, no follow-up will be required.
  Ankylosing Spondylitis Disease Activity Score (ASDAS)
Global well-being for AS patients | Day 1, no follow-up will be required.
  Bath Ankylosing Spondylitis Global score (BAS-G)
Flexibility and spinal mobility for AS patients | Day 1, no follow-up will be required.
  Bath Ankylosing Spondylitis Metrology Index (BASMI)
Chest expansion | Day 1, no follow-up will be required.
  Chest expansion will be measured circumferentially using a tape measure
Forward bending | Day 1, no follow-up will be required.
  Finger-to-Floor Distance in centimetres (cm) will be measured using a tape measure
Isometric endurance of the trunk extensor muscles | Day 1, no follow-up will be required.
  Ito test
Isometric endurance of the the trunk flexor muscles | Day 1, no follow-up will be required.
  Shirado test
Grip strength | Day 1, no follow-up will be required.
  Hand grip dynamometer (Jamar Hydraulic Hand Dynamometer)
Functional performance | Day 1, no follow-up will be required.
  50-foot walk test
Functional performance and endurance | Day 1, no follow-up will be required.
  6-min walk distance (6MWD) test

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Wilson, Principal Investigator — Trinity College Dublin, Ireland; Lolwah A Al-Rashed, Principal Investigator — Trinity College Dublin, Ireland; Finbar O'Shea, Principal Investigator — St. James's Hospital, Dublin, Ireland; Deborah Falla, Principal Investigator — University Medical Center Göttingen, Georg-August University, Göttingen, Germany; Marco Barbero, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland (SUPSI), Manno, Switzerland; Aisling Brenan, Principal Investigator — Adelaide and Meath Hospital Dublin incorporating the National Children's Hospital (Tallaght Hospital), Dublin, Ireland
Locations (3):
- Ireland (3):
  - Physiotherapy Department, Adelaide and Meath Incorporating the National Children's Hospital (Tallaght Hospital), Dublin
  - Ankylosing Spondylitis clinic, Rheumatology Department, St. James's Hospital, Dublin
  - Physiotherapy Department, St. James's Hospital, Dublin